CLINICAL TRIAL: NCT02893020
Title: National Study of the Psychological Consequences Resulting From the Practice of Invasive Therapeutic Interventions: Mixed Evaluation, Qualitative and Quantitative, of Burn Out Among Digestive Surgeons, Gastroenterologists and Radiologists
Brief Title: Emotional Experience and Burnout in Physician
Acronym: ETRE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: PHRQ14591
Record Dates: First submitted 2016-08-25; First posted 2016-09-08 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-08

CONDITIONS: Emotional Experience and Burnout in Physicians
Keywords: Emotional experience and burnout in physicians

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Recent studies have highlighted a high incidence of burnout among surgeons. The aim of this study is in particular to investigate if this is the consequence of performing surgery (i.e. invasive procedures) or whether it is related to the cultural background of surgeons.

DETAILED DESCRIPTION:
A mixed method approach (qualitative approach and quantitative approach) will be used to investigate surgeons, as well as gastroenterologists and radiologists who perform invasive procedures and gastroenterologists and radiologists who do not perform invasive procedures. The qualitative approach will rely on face-to face interviews with purposively sampled physicians of the 5 groups and will be continued until saturation. The quantitative approach will rely on a questionnaire that will be sent to physicians of the 5 groups.

ELIGIBILITY:
Inclusion Criteria:

* Digestive surgeon, Gastroenterologist, Radiologist

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Digestive surgeon, Gastroenterologist, Radiologist
Sampling Method: Non-Probability Sample
Enrollment: 3390 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
incidence of burnout | quantitative approach 27 months
  Compare the emotional experience and incidence of burnout between surgeons, gastroenterologists and radiologists

SECONDARY OUTCOMES:
physicians understanding of the Maslach Burnout Inventory (MBI) questionnaire will be reported by interview | quantitative approach 27 months
physician's emotions will be reported by interview and MBI questionnaire | quantitative approach 27 months
  concordance between the questionnaire and the interview
Correlation score depending on the specialty and professional experience | quantitative approach 27 months
  Evaluation of the MBI score over time

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Farges, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sibeoni J, Bellon-Champel L, Verneuil L, Siaugues C, Revah-Levy A, Farges O. Workplace environment around physicians' burnout: A qualitative study in French hospitals. Scand J Work Environ Health. 2021 Oct 1;47(7):521-530. doi: 10.5271/sjweh.3977. Epub 2021 Aug 7. PMID 34363393